CLINICAL TRIAL: NCT03519347
Title: Radar-A: A Phase 2 Multi-center Study to Evaluate the Safety and Tolerability of Using Point-of-Care-Guided Manipulation of Dialysate Potassium and Dialysate Bicarbonate to Prevent Hemodialysis-Associated Arrhythmias
Brief Title: Reducing Arrhythmia in Dialysis by Adjusting the Rx Electrolytes/Ultrafiltration, Study A
Acronym: RADAR-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Duke University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18-01324; R34HL140477-01 (NIH)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: End Stage Renal Disease
Keywords: arrythmia; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Potassium Removal Maximization Strategy (Experimental): Dialysate potassium will be adjusted according to the results of point of care testing in order to maximize potassium removal and avoid hyperkalemia.
  Interventions: Other: Potassium Removal Maximization; Diagnostic Test: Point of Care Testing; Device: Cardiac Monitor
- Potassium Gradient Minimization Strategy (Experimental): Dialysate potassium will be adjusted according to the results of point of care testing in order to minimize the flux of potassium.
  Interventions: Other: Potassium Gradient Minimization; Diagnostic Test: Point of Care Testing; Device: Cardiac Monitor
- Alkalosis Avoidance Strategy (Experimental): Dialysate bicarbonate concentration will be adjusted according to the results of point of care testing in order to prioritize avoiding alkalosis.
  Interventions: Other: Alkalosis Avoidance; Diagnostic Test: Point of Care Testing; Device: Cardiac Monitor
- Acidosis Avoidance Strategy (Experimental): Dialysate bicarbonate concentration will be adjusted according to the results of point of care testing in order to prioritize avoiding acidosis.
  Interventions: Other: Acidosis avoidance; Diagnostic Test: Point of Care Testing; Device: Cardiac Monitor

INTERVENTIONS:
Other: Potassium Removal Maximization — This intervention will test whether prioritizing lower potassium dialysate to reduce the incidence of hyperkalemia reduces the incidence of clinically significant arrhythmias compared to an approach minimizing intradialytic fall in serum potassium by using higher potassium dialysates to minimize serum-dialysate potassium gradients. This will be achieved by utilizing an algorithm which couples point-of-care-testing with the choice of one of two dialysate potassium concentrations (2 or 3 mEq/L) that are widely available in dialysis clinics.
  Arms: Potassium Removal Maximization Strategy
Other: Potassium Gradient Minimization — This intervention will test whether minimizing intradialytic fall in serum potassium by using higher potassium dialysates to minimize serum-dialysate potassium gradients reduces the incidence of clinically significant arrhythmias compared to an approach prioritizing lower potassium dialysate to reduce the incidence of hyperkalemia. This will be achieved by utilizing an algorithm which couples point-of-care-testing with the choice of one of two dialysate potassium concentrations (2 or 3 mEq/L) that are widely available in dialysis clinics.
  Arms: Potassium Gradient Minimization Strategy
Other: Alkalosis Avoidance — The bicarbonate (HCO3) concentration will be adjusted according to the results of point of care testing of serum chemistries and an algorithm prioritizing alkalosis avoidance by use of lower dialysate HCO3 concentrations.
  Arms: Alkalosis Avoidance Strategy
Other: Acidosis avoidance — The bicarbonate (HCO3) concentration will be adjusted according to the results of point of care testing of serum chemistries and an algorithm prioritizing acidosis avoidance by use of higher dialysate HCO3 concentrations.
  Arms: Acidosis Avoidance Strategy
Diagnostic Test: Point of Care Testing — POC testing will use the Abbott BLUE I-STAT CHEM8+ , a portable, handheld device that provides lab quality analysis within 2-3 minutes using a few drops of whole blood (≤100uL).
  Other Names: BLUE I-STAT CHEM8+
Device: Cardiac Monitor — Device is one-third of the size of a triple-A battery and is placed subcutaneously in the left chest during a brief procedure that can be done in-office under local anesthesia.
  Other Names: LINQ (Medtronic) Implantable Cardiac Loop Recorder (Carelink System)

SUMMARY:
The primary purpose of this study is to test the feasibility of trials which change the dialysate (dialysis bath prescription) of potassium and bicarbonate according to a standardized algorithm and according to the results of blood testing performed prior to each dialysis. In addition, the trial will provide estimates of the extent to which performing dialysis in this way lowers the risk of abnormal heart rhythms in people with kidney failure who are being treated with chronic hemodialysis.

DETAILED DESCRIPTION:
Within four weeks of consent, subjects will have an Implantable Loop Recorder (ILR) (Medtronic LINQ) device implanted. Subjects will be given a transmitter/charger and a Patient Care Assistant which they will be required to keep for the duration of their participation in the study. ILR tracings will be uploaded automatically and reviewed by the study team for the occurrence of clinically significant arrhythmia.

Following ILR implantation, subjects will have 1 month of standard dialysis and will crossover in random order between four month-long periods of dialysis guided by the results of the point of care testing. Whole blood will be obtained by dialysis staff and immediately tested on a point of care chemistry analyzer according to the manufacturer's protocol prior to each dialysis session. The randomized intervention periods will include algorithms that alter the potassium bath in order to a) maximize potassium removal or b) minimize potassium removal as well as a second set of algorithms that alter the bicarbonate bath in order to c) limit acidosis or d) limit alkalosis.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis therapy for end-stage renal disease
* Age 18-85 years (subjects between 18-40 years old will be required to have at least one of the following: history of congestive failure, diabetes, coronary or peripheral vascular disease, or arrhythmia)
* >30 days since dialysis initiation
* Ability to provide informed consent

Exclusion Criteria:

* Expected survival <6 monthsRenal transplant, transfer to home or peritoneal dialysis, or to non-study hemodialysis facility anticipated within 6 months
* Prisoners or cognitive disability preventing informed consent
* Pregnancy. A pregnancy test will be required for women of child bearing potential prior to enrollment. A pregnancy test will not be required for women past the age of child-bearing potential >55 years old, women with a history of surgical sterilization, or for women <55 years of age who have not had a menses within the past 12 months.
* Skin condition, immune dysfunction, history of multiple infections or other condition which increases risk of local infection with ILR placement
* Bleeding disorder or anti-coagulation that cannot be reversed for ILR placement
* Existing pacemaker, implantable monitor or defibrillator which precludes device placement
* Chronic, persistent AF. Defined as the presence of persistent AF on all available EKGs at time of recent screening.
* Hemoglobin <8 g/dL-Serum K >6.5 or <3.5 mEq/L within 30 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Charytan, MD, MSc, Principal Investigator — NYU Langone Health
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Sequence B1B2K1K2: Participants assigned to receive Alkalosis Avoidance Strategy, then Acidosis Avoidance Strategy, then Potassium Removal Maximization Strategy, then Potassium Gradient Minimization Strategy.
- Intervention Sequence B2B1K2K1: Participants assigned to receive Acidosis Avoidance Strategy, then Alkalosis Avoidance Strategy, then Potassium Gradient Minimization Strategy, then Potassium Removal Maximization Strategy.
- Intervention Sequence K1K2B1B2: Participants assigned to receive Potassium Removal Maximization Strategy, then Potassium Gradient Minimization Strategy, then Alkalosis Avoidance Strategy, then Acidosis Avoidance Strategy.
- Intervention Sequence K2K1B2B1: Participants assigned to receive Potassium Gradient Minimization Strategy, then Potassium Removal Maximization Strategy, then Acidosis Avoidance Strategy, then Alkalosis Avoidance Strategy.
Period: Baseline Observation Period
Arm/Group | Intervention Sequence B1B2K1K2 | Intervention Sequence B2B1K2K1 | Intervention Sequence K1K2B1B2 | Intervention Sequence K2K1B2B1
Started | 5 | 4 | 4 | 6
Completed | 5 | 4 | 4 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Interventional Crossover Period 1
Arm/Group | Intervention Sequence B1B2K1K2 | Intervention Sequence B2B1K2K1 | Intervention Sequence K1K2B1B2 | Intervention Sequence K2K1B2B1
Started | 5 | 4 | 4 | 6
Completed | 5 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1
Period: Interventional Crossover Period 2
Arm/Group | Intervention Sequence B1B2K1K2 | Intervention Sequence B2B1K2K1 | Intervention Sequence K1K2B1B2 | Intervention Sequence K2K1B2B1
Started | 4 (1 participant in the B1B2K1K2 experienced Death after completing the Interventional Crossover Period 1 and before starting Interventional Crossover Period 2, decreasing the number of participants who started the period from n = 5 to n = 4.) | 4 | 4 | 5
Completed | 4 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Interventional Crossover Period 3
Arm/Group | Intervention Sequence B1B2K1K2 | Intervention Sequence B2B1K2K1 | Intervention Sequence K1K2B1B2 | Intervention Sequence K2K1B2B1
Started | 3 (1 participant in the B1B2K1K2 arm experienced Death after completing the Interventional Crossover Period 2 and before starting Interventional Crossover Period 3, decreasing the number of participants who started the period from n = 4 to n = 3.) | 4 | 4 | 5
Completed | 3 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Interventional Crossover Period 4
Arm/Group | Intervention Sequence B1B2K1K2 | Intervention Sequence B2B1K2K1 | Intervention Sequence K1K2B1B2 | Intervention Sequence K2K1B2B1
Started | 3 | 4 | 3 (1 participant in the K1K2B1B2 arm experienced Death after completing Interventional Crossover Period 3 and before starting Interventional Crossover Period 4, decreasing the number of participants who started the period from n = 4 to n = 3.) | 5
Completed | 3 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Sequence B1B2K1K2 | Intervention Sequence B2B1K2K1 | Intervention Sequence K1K2B1B2 | Intervention Sequence K2K1B2B1 | Total
Number analyzed (Participants) | 5 | 4 | 4 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (13.0) | 59.7 (8.92) | 64.0 (12.8) | 54.0 (11.9) | 59.9 (11.655)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 3
  Male | 4 | 3 | 4 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 1 | 4
  Not Hispanic or Latino | 3 | 4 | 3 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 4 | 8
  White | 1 | 2 | 3 | 1 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 4 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Adherence With Proposed Interventions
Description: Adherence will be assessed as the percent of sessions in which POC testing is completed and the dialysate is adjusted according to the algorithm.
Time Frame: Up to Week 24
Measure: Mean (95% Confidence Interval); unit: Percentage of sessions
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
Number analyzed (Participants) | 17 | 16 | 16 | 17
Percentage of sessions | 88 [82 to 92] | 90 [85 to 94] | 83 [77 to 88] | 80 [74 to 85]

2. Primary Outcome: Number of Participants Enrolled Per Month
Description: Assessment of recruitment feasibility.
Time Frame: Up to Week 24
Measure: Number; unit: Patients per month
Groups:
- Overall Study Population: Overall population of participants.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 19
Patients per month | 0.7

3. Primary Outcome: Proportion of Participants Who Experienced Potassium Intervention-Specific Complications
Description: Potassium Intervention-Specific Complications are defined as either severe potassium abnormalities (potassium ≥ 6.5 or ≤ 3.0 mEq/L) or unscheduled HD or hospitalization for hyper/hypokalemia in the absence of a missed treatment.
Time Frame: Up to Week 24
Measure: Number; unit: Proportion of participants
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy
Number analyzed (Participants) | 17 | 16
Proportion of participants | 0.0062 | 0

4. Primary Outcome: Proportion of Participants Who Experience Bicarbonate Intervention-Specific Complications
Description: Bicarbonate Intervention-Specific Complications are defined as severe HCO3 abnormalities (HCO3 <20 or >32 mEq/L) or unscheduled HD or hospitalization for acid base abnormalities in the absence of a missed treatment.
Time Frame: Up to Week 24
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
Number analyzed (Participants) | 16 | 17
Proportion of participants | 0.17 [0.11 to 0.25] | 0.046 [0.02 to 0.09]

5. Primary Outcome: Mean Monthly Duration of Clinically Significant Arrhythmia (CSA)
Description: CSA will be defined on the basis of arrhythmias likely to lead to sudden cardiac arrest (SCA) or serious morbidity and mortality and will include AF, asystole ≥3 seconds, bradycardia ≤40 beats per minute lasting ≥6 seconds, and sustained VT ≥130 beats per minute lasting ≥30 seconds.
Time Frame: Up to Week 24
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
Number analyzed (Participants) | 17 | 16 | 16 | 17
Seconds | 497 (817) | 60.8 (56) | 1020 (2060) | 7950 (26000)

6. Secondary Outcome: Percent of Sessions in Which POC-Guided Dialysate Prescription Differs From Standard of Care-Guided Prescription
Description: The impact of POC testing on trial design will be measured as the percent of sessions in which the POC-guided dialysate prescription differs from a hypothetical prescription in which the choice of dialysate is based solely on the once-monthly lab (usual care).
Time Frame: Up to Week 24
Measure: Mean (Standard Deviation); unit: Percentage of sessions
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
Number analyzed (Participants) | 17 | 16 | 16 | 17
Percentage of sessions | 55.80 (49.10) | 41.20 (33.70) | 90.20 (20.10) | 88.90 (26.20)

7. Secondary Outcome: Mean Duration of Atrial Fibrillation
Time Frame: Up to Week 24
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
Number analyzed (Participants) | 17 | 16 | 16 | 17
Seconds | 1440 (0) | 120 (0) | 1170 (2180) | 189 (110)

8. Secondary Outcome: Incidence of Potentially Lethal Arrhythmias
Description: Potentially lethal arrhythmias defined as asystole, sustained VT, bradycardia for ≥6 seconds.
Time Frame: Up to Week 24
Measure: Mean (Standard Deviation); unit: Number of Potentially Lethal Arrhythmias
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
Number analyzed (Participants) | 17 | 16 | 16 | 17
Number of Potentially Lethal Arrhythmias | 2 (1.32) | 2 (1.32) | 0 (0) | 3 (1.57)

9. Secondary Outcome: Number of Screened Patients Who Are Enrolled
Description: Secondary feasibility measure to assess the size of the necessary screening pool.
Time Frame: Up to Week 24
Measure: Count of Participants; unit: Participants
Groups:
- Screening Pool: Overall pool of participants who were screened.
Arm/Group | Screening Pool
Number analyzed (Participants) | 94
Participants | 19

10. Secondary Outcome: Incidence of Hospitalization
Time Frame: Up to Week 24
Measure: Number; unit: Number of Hospitalizations
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
Number analyzed (Participants) | 17 | 16 | 16 | 17
Number of Hospitalizations | 3 | 4 | 2 | 3

11. Secondary Outcome: All-Cause Mortality
Description: Number of participants who die due to any cause.
Time Frame: Up to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
Number analyzed (Participants) | 17 | 16 | 16 | 17
Participants | 1 | 0 | 1 | 2

12. Secondary Outcome: Cardiovascular Mortality
Description: Number of participants who die due to cardiovascular-related causes.
Time Frame: Up to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
Number analyzed (Participants) | 17 | 16 | 16 | 17
Participants | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: regular investigator assessment
Arm/Group | Potassium Removal Maximization Strategy | Potassium Gradient Minimization Strategy | Alkalosis Avoidance Strategy | Acidosis Avoidance Strategy
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/16 | 1/16 | 2/17
Serious Adverse Events (participants affected / at risk) | 3/17 | 3/16 | 3/16 | 5/17
Other Adverse Events (participants affected / at risk) | 4/17 | 3/16 | 1/16 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Potassium Removal Maximization Strategy (N=17) | Potassium Gradient Minimization Strategy (N=16) | Alkalosis Avoidance Strategy (N=16) | Acidosis Avoidance Strategy (N=17)
Peripheral Angiogram (Surgical and medical procedures) | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Illeostomy closure (Surgical and medical procedures) | 0 | 1 | 0 | 0
Kidney stones (Renal and urinary disorders) | 0 | 0 | 0 | 1
Sudden visual loss (Eye disorders) | 0 | 1 | 0 | 0
Vascular access site complication (Vascular disorders) | 2 | 1 | 0 | 0
Vascular access site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Potassium Removal Maximization Strategy (N=17) | Potassium Gradient Minimization Strategy (N=16) | Alkalosis Avoidance Strategy (N=16) | Acidosis Avoidance Strategy (N=17)
Abcess (Infections and infestations) | 0 | 1 | 0 | 0
Athralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cramping (Vascular disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Kidney stones (Renal and urinary disorders) | 1 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Puncture wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular access site complication (Vascular disorders) | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT03519347/Prot_SAP_000.pdf